CLINICAL TRIAL: NCT04993469
Title: Patient Reported Outcome on Genital Sensitivity and Sexual Function After Genital Gender Affirming Surgery
Acronym: PROGAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B6702021000410
Record Dates: First submitted 2021-06-04; First posted 2021-08-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Gender Dysphoria
Keywords: Phalloplasty; Metoidioplasty; Vaginoplasty; Vulvoplasty
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Intervention Model Description: Single group assignment Single centre open label prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genital sensation and sexual functioning assessment (Experimental): Genital sensation testing with clinical assessment and self-examination questionnaire.
  Sexual functioning testing with questionnaires.
  Interventions: Diagnostic Test: Semmes-Weinstein monofilament testing and questionnaires

INTERVENTIONS:
Diagnostic Test: Semmes-Weinstein monofilament testing and questionnaires — Semmes-Weinstein test for the assessment of genital sensation Battery of questionnaires assessing sexual function, voiding function, quality of life and patient satisfaction

SUMMARY:
For genital gender affirming surgery, it remains unclear to what extent genital sensitivity might be expected and what the impact of this might be on sexual functioning.

DETAILED DESCRIPTION:
Gender dysphoria refers to an inner mental unrest resulting from an incongruity between the assigned biological sex and the mentally experienced sex. The generally accepted treatment for gender dysphoria aims to bring a person's physical characteristics in line with his or her perceived gender identity. This gender-affirming treatment consists of a combination of psychological counselling, hormonal therapy and, if desired, genital gender-affirming surgery. This involves the removal of the biological reproductive organs and in some cases (part of) the biological sex organs. These can be replaced by surrogate sex organs of the desired sex while maintaining urological and sexual function. In transgender women, this is achieved with vulvoplasty or vaginoplasty, while in transgender men, metoidioplasty or phalloplasty is performed.

While urological functioning is an extensively studied topic in transgender patients after genital gender confirmation surgery, sexual functioning is often considered of secondary importance, even though it is one of the goals of gender confirmation surgery. In the transgender man, a phalloplasty is performed using microsurgical techniques that allow the nerves of the donor flap (usually from the forearm or upper leg) to be connected to the genital and inguinal nerves. In metoidioplasty, the clitoris is preserved and forms the base of a micro-penis. In the transgender woman, the glans penis is partially preserved to create a clitoris. The purpose of this is to achieve maximum sensitivity of the genital area.

There are few reports in the literature demonstrating sensory recovery in these extensively operated body parts, let alone what the added value on sexual functioning might be as a result of this recovery of genital sensitivity. At Ghent University Hospital, we now have more than 30 years' experience with such operations and have shared this experience in an almost entirely retrospective manner in various publications to date. However, in order to address the bias associated with retrospective research, this study aims to prospectively and observationally collect data on these patients who are counseled in a pathway for gender dysphoria. This study will include all patients - after informed consent - and will collect specific data on surgical outcome (complications after surgery, duration of surgery, type of surgery) and functional outcome (tailored questionnaires for patients undergoing such a treatment with questions on urination, erections, sexual experience, quality of life, patient satisfaction and genital sensitivity) for each of these various surgical options. These outcomes will be verified at follow-up moments (after 3 months, 6 months, 12 months and 24 months). Specifically for the component on genital sensitivity, we plan to follow up patients 3-monthly by means of a Semmes-Weinstein monofilament test of the genital region up to 24 months postoperatively. The aim of this study is therefore to use this prospectively collected data to truthfully map our experience, to be critical, to reflect and optimize our daily clinical practice in the interest of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written informed consent according to the rules of Good Clinical Practice (Declaration of Helsinki) and national regulations
* Patient age ≥ 18 years
* Transgender male, female of gender non-conforming patient with diagnosed gender dysphoria and the specific wish to undergo genital gender affirming surgery
* Fit for operation, based on the surgeon's expert opinion
* Patient is able and willing to attend the follow-up consultations

Exclusion Criteria:

* Absence of signed written informed consent and thus a patient unwilling to participate.
* Patient age < 18 years
* Cisgender patients
* Patients unfit for operation
* Patient declares that it will be impossible for him to attend the follow-up consultations

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is specific to patients with gender dysphoria who wish to undergo genital gender affirming surgery.
Enrollment: 200 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in genital sensitivity pattern at 24 months | Baseline function test, followed by reassessment at 3, 6, 9, 12, 15, 18, 21 and 24 months of follow-up
  Mapping of pressure thresholds of Semmes-Weinstein monofilaments in pre-defined areas of the neo-genital area

SECONDARY OUTCOMES:
Change in postoperative sexual function | Baseline questionnaire, followed by reassessment at 12 and 24 months of follow-up
  Assessed with Male Sexual Health Questionnaire/Female Sexual Function Index questionnaires (MSHQ/FSFI) with added questions specifically on penetrative sexual activity
Change in self-assessment of genital anatomy and genital sensitivity | Baseline questionnaire, followed by reassessment at 3, 6, 9, 12, 15, 18, 21 and 24 months of follow-up
  Assessed with Self-Assessment of Genital Anatomy and Sexual Function (Male and Female) questionnaires (SAGASF-M/SAGASF-F)
Change in voiding function | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed with International Consultation on Incontinence Questionnaire on Male and Female Lower Urinary Tract Symptoms (ICIQ-MLUTS/ICIQ-FLUTS)
Change in urinary continence | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed with International Consultation on Incontinence Questionnaire on Urge Incontinence short form questionnaire (ICIQ-UI SF)
Change in maximum flow rate | Uroflowmetry at baseline, followed by uroflowmetry at 3, 6, 12 and 24 months of follow-up
  Assessed by uroflowmetry (Qmax)
Change in satisfaction with life by Likert and VAS scales | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed with Satisfaction with life scale (SWLS) questionnaire
Change in satisfaction with life by Likert and VAS scales | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed with Subjective happiness scale (SHS) questionnaire
Change in quality of life assessed by Likert scales. | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed by the EuroQol questionnaire EQ-5D-3L.
Change in quality of life assessed by VAS scale. | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed by the EuroQol questionnaire EQ-VAS (0-100)
Subjective patient satisfaction with surgical and functional outcome assessed by Likert scales. | Assessed at 12 and 24 months of follow-up
  Assessed with seven subjective patient satisfaction questions on different surgical and functional outcomes aspects using Likert scales
Patient motivations for surgery and extent to which these expectations were met as a result of the operation assessed by VAS scales | Baseline questions, followed by reassessed at 12 and 24 months of follow-up
  Assessed with fourteen motivational questions using VAS scales (0-100)
Postoperative complication rate | Within 90 days postoperatively
  Categorized according to Clavien-Dindo classification system

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No